CLINICAL TRIAL: NCT04895215
Title: A Randomized, Double-blind, Placebo-controlled Study of the Efficacy, Safety, and Tolerability of AB-2004 in an Autism Spectrum Disorder Population
Brief Title: AB-2004 in Treatment of Irritability Associated With Autism Spectrum Disorder (ASD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertero Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AXL-2004-002
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Autism Spectrum Disorder (ASD)
Keywords: Irritability; Anxiety
MeSH Terms: conditions — Autism Spectrum Disorder; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Double Blind, Randomized, Placebo Controlled
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AB-2004 (Experimental)
  Interventions: Drug: AB-2004
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AB-2004 — Taken 3 times daily with food
  Arms: AB-2004
Drug: Placebo — Take 3 times daily with food
  Arms: Placebo

SUMMARY:
The purpose of this study is to establish the potential benefits, safety, and tolerability of AB-2004 in participants with irritability associated with autism spectrum disorder.

ELIGIBILITY:
Key Inclusion Criteria:

* Clinically diagnosed, documented ASD (Diagnostic and Statistical Manual of Mental Disorders [DSM-5] criteria)
* Aberrant Behavior Checklist - Irritability (ABC-I) score ≥18 at the Screening Period
* Clinical Global Impression - Severity (CGI-S) scale score ≥4 at the Screening Period

Key Exclusion Criteria:

* Use of an oral, injected, or inhaled antibiotic within 30 days prior to screening. Prophylactic oral antibiotic use of no more than 1 dose will be permitted
* Current use of an oral controlled or extended-release medication
* Have a comorbid major psychiatric condition (eg, schizophrenia or bipolar disorder) at screening that in the opinion of the Investigator may interfere with the subject's ability to complete study procedures/comply with study requirements
* Current use of antipsychotics (eg, aripiprazole or risperidone)

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 156 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
The mean change in the ABC-I score (Irritability) from Baseline to Week 8 for AB-2004 | From baseline to Week 8 visit

SECONDARY OUTCOMES:
The mean change in the Clinical Global Impression-Severity (CGI-S) from Baseline to Week 8 for AB-2004 High Dose and AB-2004 Low Dose | From baseline to Week 8 visit
Number of participants who reported treatment emergent adverse events (TEAEs) | From baseline to Week 8 visit

CONTACTS AND LOCATIONS:
Locations (24):
- United States (18):
  - Harmonex Neuroscience Research, Dothan, Alabama
  - Southwestern Autism Research and Resource Center, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - Cortica Marin, San Rafael, California
  - Cortica Westlake, Westlake Village, California
  - IMMUNOe Research Centers, Centennial, Colorado
  - Yale University, New Haven, Connecticut
  - CNS Solutions, Jacksonville, Florida
  - CNS Solutions, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Baber Research, Naperville, Illinois
  - University of Missouri, Thompson Center for Autism and Neurodevelopmental Disorders, Columbia, Missouri
  - Clinical Research of Southern Nevada, Las Vegas, Nevada
  - Spectrum Neuroscience and Treatment Institute, New York, New York
  - Nathan S. Kline Institute for Psychiatric Research, Orangeburg, New York
  - Ohio State University, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Relaro Medical Trials, Dallas, Texas
- Australia (5):
  - Brain Mind Centre, Sydney, New South Wales
  - Westmead Children's Hospital, Sydney, New South Wales
  - Children's Health Queensland Hospital, South Brisbane, Queensland
  - Monash Kids Research, Clayton, Victoria
  - Murdoch Children's Research Institute, Parkville, Victoria
- Optimal Clinical Trials, Grafton, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No